CLINICAL TRIAL: NCT00292747
Title: Comparison of the Efficacy and Tolerability of Drotaverine 80 mg, Ibuprofen 400 mg and Their Combination in a Calendar Packaging for the Treatment of Primary and Secondary Dysmenorrhoea
Brief Title: Drotaverine in Dysmenorrhoea Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: early termination due to loss of interest and low enrollment of patient
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_9134
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — drotaverin; Ibuprofen

ARMS (3):
- drotaverine + Ibuprofen placebo (Experimental): Drotaverine 80 mg plus ibuprofen placebo orally
  Interventions: Drug: Drotaverine; Drug: Ibuprofen Placebo
- Drotaverine placebo + ibuprofen (Active Comparator): Drotaverine placebo plus ibuprofen 400 mg orally
  Interventions: Drug: Drotaverine Placebo; Drug: Ibuprofen
- Drotaverine + ibuprofen (Active Comparator): Drotaverine 80 mg plus ibuprofen 400 mg orally
  Interventions: Drug: Drotaverine; Drug: Ibuprofen

INTERVENTIONS:
Drug: Drotaverine
  Other Names: Z0124
  Arms: Drotaverine + ibuprofen; drotaverine + Ibuprofen placebo
Drug: Drotaverine Placebo
  Arms: Drotaverine placebo + ibuprofen
Drug: Ibuprofen
  Arms: Drotaverine + ibuprofen; Drotaverine placebo + ibuprofen
Drug: Ibuprofen Placebo
  Arms: drotaverine + Ibuprofen placebo

SUMMARY:
The aim of the study is to show that the combination of drotaverine 80mg and ibuprofen 400 mg is more effective and as well-tolerated as ibuprofen 400 mg or drotaverine 80 mg administered alone, in the treatment of primary and secondary dysmenorrhoea.

ELIGIBILITY:
Inclusion Criteria:

* History of at least 6 months of dysmenorrhea, with presence of moderate to severe pain in each of the last 3 cycles
* With regular menstrual cycles (25-35 days)
* Using an adequate barrier contraception method (except for virgins)

Exclusion Criteria:

* Evidence of clinically relevant gynecological, cardiovascular, hematologic, hepatic, gastrointestinal, renal, pulmonary, endocrinologic, neurologic or psychiatric disease, based on a clinical assessment and routine laboratory investigations
* Proven hypersensitivity to drotaverine hydrochloride or ibuprofen or proven intolerance to lactose
* Any described contraindication to either drotaverine hydrochloride or ibuprofen (see Summary of Product Characteristics)
* Oestro-progestative contraception within the last 2 months
* Regular use of sedative, hypnotics, tranquillizers or any other addictive agents
* History or evidence of acute or chronic alcohol abuse
* Heavy smoking (> 10 cigarettes/day)
* Need of a permanent treatment with other antispasmodics and/or analgesic agents during the trial
* Lactation
* Pregnancy
* Participation in another clinical trial in the last 3 months prior to the start of this study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 480
Dates: Start 2005-05-25 (Actual); Primary Completion 2006-02-28 (Actual); Study Completion 2006-02-28 (Actual)

PRIMARY OUTCOMES:
Reponse rate in each treatment arm: proportion of patients having pain intensity score 0 or 1 at hour 2 after the first drug intake.

CONTACTS AND LOCATIONS:
Overall Officials: László Erős, MD, Study Director — Sanofi-aventis, Hungary
Locations (1):
- Sanofi-Aventis, Budapest, Hungary